CLINICAL TRIAL: NCT07083089
Title: Phenotyping of Audition in Patients With Early Stage of Neurodegenerative Disorders (Alzheimer and Parkinson' Diseases)
Brief Title: Early Stage of Alzheimer's and Parkinson's Diseases, HearIng Relevance (SAPHIR)
Acronym: SAPHIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cilcare SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024-A01578-39
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment (MCI) Amnestic; Parkinson Disease (PD); Healthy Participants
Keywords: hearing phenotype; audiometry; speech-in-noise intelligibility; electrophysiology
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Eligibile patients are included and subject to a thorough hearing assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): Control population
  Interventions: Other: Thorough Hearing assessment
- Amnestic MCI Group (Experimental): Patients with amnestic mild cognitive impairment
  Interventions: Other: Thorough Hearing assessment
- Parkinson Group (Experimental): Patient with parkinson's disease
  Interventions: Other: Thorough Hearing assessment

INTERVENTIONS:
Other: Thorough Hearing assessment — Otoscopy Tympanometry Tonal audiometry (air and bone conduction) Vocal audiometry (in silence and in noise) Distorsion Products of OtoAcoustic Emissions (DPOAE) Middle Ear Muscle Reflex (MEMR) Auditory Brainstem Response (ABR) Electrocochleography (EcochG)

SUMMARY:
The study aims to phenotype hearing in patients with early stage of neurodegenerative disorders to explore the prevalence of various hearing disorders in comparison to a control population. Specific focus is made on patients with speech-in-noise intelligibiltiy deficit despite normal tonal audiograms referred to as hidden hearing loss, with potential identification of associated biomarkers.

DETAILED DESCRIPTION:
A wide battery of subjective and objective hearing tests is performed on the subjects including tonal and vocal audiometry (in silence and in noise), DPOAE, acoustic reflex and electrophysiology recordings (auditory brainstem response, electrocochleography). Hearing tests are correlated to collected disease parameters and blood markers.

ELIGIBILITY:
Inclusion Criteria: All subjects

1. Man or woman aged between 50 and 85 years old at baseline.
2. Fluent in French (native language)
3. Be considered as reliable and capable of adhering to the protocol, according to the judgment of the investigator (understanding of the information included in the protocol, and requests to realize the investigations, good general health and able to move around).
4. Affiliated to Public Health Insurance (Sécurité Sociale)
5. Signed and dated informed consent form.

For amnestic MCI:

Diagnosis of amnestic MCI, according to international diagnosis criteria (NIA-AA, 2011) with MoCA≥23 or MMSE>24.Patients must exhibit predominantly cognitive impairments in episodic memory, defined by a score on the RL/RI 16-item test with a free recall score of less than 18/48 and a total recall score of less than 40/48.

For Parkinson Patients:

Established clinical diagnosis of Parkinson's disease according to Postuma et al. 2015 with bradykinesia associated with resting tremor or rigidity, no exclusion criteria or red flag with MOCA ≥23.

For controls:

No diagnosis of neurological disease such as Parkinson's disease or MCI associated or not with Alzheimer's disease Displays normal cognitive status with a MoCA score ≥ 26.

Non-inclusion criteria:

1. Known hearing pathologies leading to conductive hearing loss (otosclerosis, a diagnosed pathology of the ear canal, tympanic membrane, ossicles or 3rd window), otitis, congenital deafness or sensorineural hearing loss associated to Menière's disease.
2. Psychiatric diseases other than neurodegenerative etiology
3. Neurological or neurovascular disorders (Stroke, epilepsy, dementia)
4. Motor complications that could interfere with audiological assessment
5. Known Diagnosis of type 2 diabetes
6. Alcohol or drug addiction
7. Cochlear implant
8. Known ototoxic drug therapy:

   1. Antibiotics: Aminosides IV, macrolides, tetracyclines in the last 15 days prior to inclusion
   2. Antipaludic drugs: quinine, hydroxychloroquine, chloroquine in the last 15 days prior to inclusion
   3. Platinum-based chemotherapy at any time prior to inclusion.
   4. Loop diuretics: furosemide (max oral dose of ≤60mg/day) at inclusion and during the study.
   5. Salicylate derivatives at high dose (Kardegic allowed at dose ≤320mg/day) at inclusion and during the study.
9. History of otological surgical act.
10. On-going pregnancy or breast-feeding.
11. Adults protected by law: in vulnerable social situations or unable to express consent.
12. Under another protocol that may interfere with the analysis of the results.

Exclusion Criteria:

Patients will be excluded from the study if one or more of the following criteria are applicable during visit 2:

1. Abnormal otoscopy as defined by less than 90% of the tympanic membrane visible (cerumen ear plug, ear drum perforation, …)
2. Conductive hearing loss defined by an air-bone threshold gap of 10 dB or greater based on the average of frequencies 0.5, 1, 2, and 4 kHz, and abnormal hearing thresholds (greater than 20 dB HL) for these frequencies.
3. Abnormal tympanogram (other type than A)
4. Asymmetric hearing loss: more than 15 dB difference in the pure-tone average (PTA) air conduction (for MCI patients and control group only)
5. Single-sided deafness (SSD)
6. Cophosis (PTAv > 120 dB)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hidden hearing loss | within one month from inclusion
  Percentage of population in each group that displays normal audiometric thresholds (0.5-4kHz) and impaired speech-in-noise intelligibility

SECONDARY OUTCOMES:
Prevalence of sensorineural hearing loss | within one month from inclusion
  Percentage of patients in each group with elevated hearing thresholds (0.5-4kHz)
Grade of sensorineural hearing loss | within one month from inclusion
  As defined by BIAP criteria : ]20-40 dB nHL] = mild ; ]40 - 55] = moderate ; ]55 - 70] = moderately severe ; ]70 - 90] = severe ; ]90 - 120] = profound ;

OTHER OUTCOMES:
Explore auditory signatures in neurodegenerative disease patients | one month from inclusion
  Determine combination of auditory results that could be discriminatory of patient population versus control group
Identify potential biomarkers of cochlear synaptopathy | one month from inclusion
  correlations between specific auditory findings and disease parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu SCHUE, PhD, Study Director — Cilcare SAS
Locations (4):
- France (4):
  - CHU Gui de Chauliac, Montpellier
  - CHU Nice, Nice
  - CHU Carémeau, Nîmes
  - Hospices Civils de Lyon, Hôpital des Charpennes, Villeurbanne

IPD SHARING:
Plan to Share IPD: No